CLINICAL TRIAL: NCT03266185
Title: Prospective, Multi-centre Trial to Evaluate Effectiveness of 45-min and 20-min Post-infusion Cooling Time for Patients Treated With Scalp Cooling to Prevent Paclitaxel-induced Alopecia
Brief Title: Shorter Scalp Cooling Time in Paclitaxel
Acronym: COP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.R. Kroep, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL61964.058.17
Record Dates: First submitted 2017-08-26; First posted 2017-08-30 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Neoplasm Malignant; Breast Cancer; Ovarian Cancer
Keywords: paclitaxel-containing chemotherapy
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 45-minutes (Experimental): 45-minutes post-infusion cooling time
  Interventions: Other: Shorter PICT
- 20-minutes (Experimental): 20-minutes post-infusion cooling time
  Interventions: Other: Shorter PICT
- No scalp cooling (No Intervention): Patients who decline scalp cooling will be included as a control group to determine the incidence of paclitaxel-induced alopecia

INTERVENTIONS:
Other: Shorter PICT — Shorter post-infusion cooling time
  Arms: 20-minutes; 45-minutes

SUMMARY:
Chemotherapy-induced alopecia (CIA) is one of the most distressing side effects for patients. Scalp cooling can prevent or minimise CIA in approximately half of all patients, depending on many factors, e.g. type and dosage of chemotherapy. High rates of success are seen in patients treated with taxanes, up to 80-90%. Previous research has shown comparable results of scalp cooling in docetaxel-treated patients when shortening the post-infusion cooling time (PICT) from the initial standard of 90 minutes to 45- and 20 minutes. A shorter PICT is an advantage for both the patient, who can spend less time in the hospital, as well for the logistics at oncological departments. Paclitaxel and docetaxel are both classical taxanes, that share similar mechanisms of action and have comparable plasma terminal half-life times, therefore it seems plausible that the PICT can be shortened for paclitaxel-treated patients as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving weekly-administered paclitaxel-containing chemotherapy (minimal 3 planned administrations) in a dose of 80-90 mg/m2 Paclitaxel monotherapy, Paclitaxel in combination with carboplatin, Paclitaxel in combination with monoclonal antibodies: Bevacizumab or Trastuzumab
* Age ≥ 18 years
* WHO performance status 0-2
* Survival expectation must be > 3 months
* Written informed consent according to the local Ethics Committee requirements

Exclusion Criteria:

* Treatment with paclitaxel in sequential schemes with other alopecia inducing agents such as paclitaxel monotherapy after adriamycin, cyclophosphamide (AC) or paclitaxel monotherapy after 5-fluouracil, epirubicin, cyclophosphamide (FEC) treatment
* Alopecia before the start of the study
* Rare cold-related disorders: Cold sensitivity, Cold agglutinin disease, Cryoglobulinaemia, Cryofibrinogenaemia, Cold posttraumatic dystrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of scalp cooling in patients treated with paclitaxel-containing chemotherapy with a 45- and 20-minutes post-infusion cooling time, defined by the patient's self-determined need to wear a wig or other head covering | up to 52 weeks

SECONDARY OUTCOMES:
To determine the degree of chemotherapy-induced alopecia (CIA), assessed with the DEAN scale for assessment of hair loss | up to 52 weeks
To determine the grade of chemotherapy-induced alopecia (CIA), according to NCI-CTCAEv4.03 | up to 52 weeks
To determine the tolerance of scalp cooling, assessed by a (self-adapted) visual analogue scale (VAS) | up to 52 weeks
To determine the added value of scalp cooling for weekly paclitaxel; what is the incidence of severe alopecia with and without scalp cooling | up to 52 weeks
Assessing the amount of distress experienced by CIA in patients, assessed with the chemotherapy-induced alopecia distress scale (CADS) | up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- LUMC, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lugtenberg RT, van den Hurk CJG, Smorenburg CH, Mosch L, Houtsma D, Deursen MAGDH, Kaptein AA, Gelderblom H, Kroep JR. Comparable effectiveness of 45- and 20-min post-infusion scalp cooling time in preventing paclitaxel-induced alopecia - a randomized controlled trial. Support Care Cancer. 2022 Aug;30(8):6641-6648. doi: 10.1007/s00520-022-07090-7. Epub 2022 May 2. PMID 35501515